CLINICAL TRIAL: NCT04145778
Title: Evaluation of the Muscular FORCE in the Upper Limbs of Patients Presenting a Thoracic Outlet Syndrome : Monocentric Case-control Study
Brief Title: Evaluation of the Muscular FORCE in the Upper Limbs of Patients Presenting a Thoracic Outlet Syndrome
Acronym: EFORD
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0387
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Thoracic Outlet Syndrome
MeSH Terms: conditions — Thoracic Outlet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient
  Interventions: Other: 6-minute walk test
- Control
  Interventions: Other: 6-minute walk test

INTERVENTIONS:
Other: 6-minute walk test — The 6-minute walk test is performed as part of routine practice for patients with BMDS to assess patients' overall endurance. In order to compare patients' global endurance with controls, this walking test will also be offered to 50 of the healthy subjects already recruited in the study.

SUMMARY:
The thoracic outlet syndrome is a rare but debilitating pathology, responsible for upper limb pain. Its frequency is probably underestimated because of diagnostic difficulties. This syndrome encompasses several entities including compressions of neurological, venous or arterial origin. In addition to pain, the majority of patients report fatigability and loss of strength in the upper limbs. However, the quantification of this loss of strength and fatigability has hardly been studied.

In addition, the rehabilitation treatment is the first-line treatment of this pathology. It most often includes a muscle building phase.

In this project, we would like to evaluate the proximal and distal force of patients presenting a thoracic outlet syndrome by comparing them to a population free from any pathology in the upper limbs. This evaluation would involve an isokinetic strength analysis of shoulder rotators at the proximal level, using an isokinetic dynamometer. At the distal level, the evaluation would be done using force clamps.Similarly, performing a 6-minute walk test will assess whether there is a difference between patients and controls, which may also impact endurance in addition to the pathology.

In a second step, we will also be able to evaluate the effects of the reeducation on the strength and the muscular fatigability of the patients presenting a thoracic outlet syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Rehabilitative management of an thoracic outlet syndrome in the physical and rehabilitation department of Nantes University Hospital
* Having given their consent by non-oral opposition.
* Affiliated to a social security scheme

Exclusion Criteria:

* Mineurs
* Majeurs under tutorship, curatorship or safeguard of justice
* Pregnant or lactating women, protected persons
* Patients with other pathology of the upper limb or shoulder (osteoarthritis, tendinopathies, amputation, ...).
* Patients with non-stabilized pathologies, heart, respiratory, metabolic or neurological conditions
* Associated pathology able to interfere with carrying out assessments

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients with an thoracic outlet syndrome will be needed, which corresponds to the annual recruitment in this care within the department of the University Hospital of Nantes.
  Patients will be included during their usual management of rehabilitation at the center.
  50 healthy subjects will be included, in order to have a patient for a healthy subject. We will call on the staff and student volunteers of the rehabilitation center we will match on age, sex and weight.
  For both groups, we will only use major topics that do not benefit from any legal protection measures
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-08-03 (Estimated); Study Completion 2024-12-03 (Estimated)

PRIMARY OUTCOMES:
Comparing proximal force between patients with thoracic outlet syndrome and healthy subjects | 1 year
  Isokinetic evaluation of the internal shoulder rotators
Comparing distal force between patients with thoracic outlet syndrome and healthy subjects | 1 year
  Isokinetic evaluation of the external shoulder rotators

SECONDARY OUTCOMES:
Muscular fatigue in patients with thoracic outlet syndrome | 1 year
  Isokinetic evaluation of internal and external shoulder rotator fatigue at 180 ° / s
Evaluation of the effects in terms of strength of rehabilitation | 1 year
  Isokinetic evaluation of rotators in strength
Evaluation of the effects in terms of fatigue of rehabilitation | 1 year
  Isokinetic evaluation of rotators in fatigue
Impact on pain | 1 year
  Visual analogue pain scale (from 0 to 10: 0 absence of pain, 10 maximum pain imaginable)
Evolution of cardiorespiratory performance | 1 month
  Evalution of changes in cardiorespiratory performance using a 6-minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Alban FOUASSON-CHAILLOUX, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided